CLINICAL TRIAL: NCT02292927
Title: Maximising Recovery to Health Through Trimodal (Bio Psycho Social) Prehabilitation for Aneurysm Surgery Study
Brief Title: Trimodal Prehabilitation for Aneurysm Surgery Study
Acronym: T-PASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14/LO/1368
Record Dates: First submitted 2014-11-06; First posted 2014-11-18 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-05

CONDITIONS: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-intervention (No Intervention): Patients treated as standard before intervention
- Post-intervention arm = Prehabilitation (Active Comparator): Introduction of rehabilitation program
  Interventions: Behavioral: Post-intervention arm = Prehabilitation

INTERVENTIONS:
Behavioral: Post-intervention arm = Prehabilitation — Introduction of a physical exercise training programme, psychological counselling and smoking cessation advice
  Arms: Post-intervention arm = Prehabilitation

SUMMARY:
DESIGN: Single-centre, feasibility study AIMS: The aim of this study is to evaluate the acceptability and pre-operative impact on functional capacity of a trimodal prehabilitation program in a cohort of patients undergoing aneurysm repair.

This will enable the design (feasibility and power) of a large scale Randomised Controlled Trial.

Expected outcomes

* The potential number of patients who would benefit, the compliance and acceptability of a pre-operative prehabilitation programme will be calculated.
* Preoperatively, expected at 6-weeks, the change in physical fitness of patients (assessed by the physical function section of SF-36 and measured with peak flow/6-minute walk testing) during the pre-operative phase will be assessed in both groups.
* The effects on quality of life, anxiety and depression on each study participant will be assessed immediately pre-op, expected at 6-weeks.
* The number of patients who are able to reduce or cease smoking will be reported during the pre-op phase (expected at 6 weeks), as will length of hospital stay after aortic surgery, expected at 6-8 weeks.

POPULATION: Patients undergoing planned elective aortic surgery procedures

ELIGIBILITY: Adult patients (over 18 years) undergoing elective open and endovascular aneurysm repair with capacity to consent and physical fitness to undergo an pre-operative exercise programme DURATION: 1 year from 1st June 2014

DETAILED DESCRIPTION:
Proposed intervention - The introduction of a biopsychosocial intervention before surgery. The physical exercise programme will be a prescribed exercise training twice per week which will be supported by a physical therapist and vascular nurse specialist. A trained clinical psychologist will also deliver a brief psychological intervention based on cognitive behavioural therapy (CBT) techniques in two sessions to modify illness, surgical preparation and rehabilitation beliefs. Lastly patients will be counselled and referred to smoking cessation services as appropriate by the vascular nurse specialist.

Baseline information will include patient demographics and medical history, quality of life assessment using SF-36 forms, hospital anxiety and depression scale (HADS) and exercise testing by a standardised 6-minute walk test Information immediately pre-operatively will be collected to include a repeat assessment of physical function with a 6-minute walk test, SF-36 assessment and HADS scores. Smoking cessation rate will be collected.

A pre and post-intervention group will be studied over a 1-year period. We will report on the eligibility, acceptability and pre-operative effect of this trimodal rehabilitation programme.

AIM AND EXPECTED IMPACT

This is a non-randomised pre-post intervention pilot study to understand the acceptability and pre-operative effects of a combined physical, psychological and social prehabilitation package in patients undergoing aneurysm repair. This will enable the design (feasibility and power) of a large scale Randomised Controlled Trial.

Our hypotheses include:

* The introduction of a prehabilitation programme will be acceptable to the majority of patients undergoing aneurysm surgery
* A physical pre-operative exercise programme will increase physical fitness before surgery
* A psychological intervention based on cognitive behaviour therapy techniques will reduce anxiety before surgery and prepare patients better for their post-operative recovery
* The introduction of psycho-social counselling for smoking cessation will encourage more patients to give up smoking pre-operatively

PARTICIPANT ENTRY: PATIENTS

PRE-REGISTRATION EVALUATIONS The research team will identify eligible patients for recruitment into the study via clinic lists, multidisciplinary meetings and referral letters before the patient attends their clinic appointment. Only adult patients undergoing aortic surgery will be selected. Patient information leaflets will be given to selected patients and patients will be given the opportunity to read them and ask questions before deciding whether or not to participate.

INCLUSION CRITERIA

* Adult patients (>18 years old) undergoing aortic aneurysm repair.
* Ability to comprehend and retain instructions regarding self-training
* Physical fitness allowing participation in an exercise programme.

EXCLUSION CRITERIA

* Minors (<18 years old)
* Adult patients who do not have capacity to consent.
* Emergency or urgent procedures who will not have a necessary 6 week lead in time until operation.

WITHDRAWRAL CRITERIA The patient will be made aware that they may withdraw from the study at any time without providing a reason; their care and treatment will not be affected

STUDY DESIGN The acceptability of this programme will be studied and the pre-operative impact on functional capacity will be assessed in a comparator (pre-intervention) and post-intervention group.

Patients

Patients from Imperial College Healthcare NHS Trust Vascular Unit undergoing aortic aneurysm repair will be recruited.

Study Protocol

Our current vascular pre-operative assessment service is an established nurse led service, run by a dedicated aortic clinical nurse specialist. The prehabilitation would run in conjunction with the current pre-operative screening measures currently in place - which include dobutamine stress echocardiography, renal assessment and pulmonary function tests.

-Phase 1 - Comparator (pre-intervention) evaluation

Patients undergoing present standard of care - i.e. standard work-up for aneurysm repair without nurse-led prehabilitation strategy, who meet inclusion and exclusion criteria will be given a patient information leaflet, informed they are in the pre-intervention group and consented for inclusion in the study as detailed above.

At the baseline appointment, on the same day as work-up tests, information will be collected on standardised data collection sheets to include:

* Patient demographics and medical history
* Baseline Quality of Life assessment using SF-36 forms
* Hospital anxiety and depression scale (HADS).
* Exercise testing by a standardised 6-minute walk test
* Peak Expiratory Flow Rate (PEFR)

Information immediately pre-operatively will be collected the day before operation (our standard admission is the day before) to include a repeat assessment of physical function with a 6-minute walk test, Peak Expiratory Flow Rate (PEFR), SF-36 assessment and HADS scores. Smoking cessation rate over the pre-operative period will be collected. The aneurysm repair will proceed as standard of care, and will be unchanged from standard practice.

-Phase 2 - Intervention

Proposed intervention - The introduction of a biopsychosocial intervention before surgery. The physical exercise programme will be prescribed exercise training twice per week which will be supported by our vascular nurse specialist, previously shown to have a small effect on length of stay in cardiac patients [12].

A trained specialist (a registered psychologist) will also deliver a brief psychological intervention based on cognitive behavioral therapy (CBT) techniques in two sessions to modify illness, surgical preparation and rehabilitation beliefs. This psychological intervention has been shown to be effective in encouraging claudicants to initiate and continue exercise training [13].

Lastly patients will be counselled and referred to smoking cessation services as appropriate.

Phase 2 protocol - During an initial set-up phase comprehensive information booklets will be developed to instruct the patient on these three modes of prehabilitation.

Patients who are eligible for the study will be approached in the same way as patients studied in the comparator group. At the baseline study visit, the same baseline information will be collected as for the comparator group i.e.:

At the baseline appointment, on the same day as work-up tests, information will be collected on standardised data collection sheets to include:

* Patient demographics and medical history
* Baseline Quality of Life assessment using SF-36 forms
* Hospital anxiety and depression scale (HADS).
* Exercise testing by a standardised 6-minute walk test
* Peak Expiratory Flow Rate (PEFR)

In addition patients will receive:

* Information booklets
* Physical exercise plan, run-through and explanations.
* Psychological therapy on this day or a mutually convenient day for patient and therapist.
* Counselling by the nurse specialist and referral for smoking cessation

Patients will receive a telephone follow-up with the nurse specialist at week 2 and week 4 to evaluate progress and to encourage compliance with the programme. Between weeks 5-6 the patient will have a further session with the clinical psychologist, just prior to admission for treatment, to prepare them for their impending hospitalisation.

Again, information immediately pre-operatively will be collected to include a repeat assessment of physical function with a 6-minute walk test, Peak Expiratory Flow Rate (PEFR), SF-36 assessment and HADS score. In addition, patients will be asked to fill out a questionnaire assessing compliance with and acceptability of the prehabilitation programme. Smoking cessation rate will be collected.

Data Collection

The following demographic data will be recorded on standardised data collection forms for each patient, collected from patient records and the patient interviews:

* Inclusion and exclusion criteria
* Medical history/risk factors
* ASA classification
* Planned operative procedure details
* Physical status using functional capacity, measured in metabolic equivalents (METs), with a Duke Activity Status Index (score of less than 4 indicates poor physical function).

Functional capacity may be usually expressed in metabolic equivalents (METs), where one MET is defined as the oxygen consumption of a 70-kg man at rest. Greater than 7 METs of activity tolerance is considered excellent, whereas less than 4 METs is considered poor activity tolerance.

The Duke Activity Status Index suggests questions that correlate with MET levels; for example, walking on level ground at about 4 miles per hour or carrying a bag of groceries up a flight of stairs expends approximately 4 METs of activity. This system is used by the Cleveland clinic for pre-operative cardiac evaluation. It allows a pre-operative assessment of physical function to assess predicted ability to cope at home after surgery. A brief, self-completed questionnaire (Appendix 1) can provide a standardized assessment of functional status that correlates well with an objective measure of maximal exercise capacity [14].

Post-operative data will be collected for patients in order to plan for a further study based on reducing length of stay.

* Inpatient complications: grade and details using standardised data collection sheets
* Length of stay
* HDU/ITU use
* Mortality

At base line visit and prior to operation each patient will be assessed using:

* Baseline Quality of Life assessment using SF-36 forms
* Hospital anxiety and depression scale (HADS).
* Exercise testing by a standardised 6-minute walk test
* Peak Expiratory Flow Rate (PEFR)

An event log will be recorded for each patient throughout the study period.

Patients undergoing intervention will be asked to complete a short questionnaire on compliance and acceptability of the prehabilitation programme.

ANALYSIS Completed data collection sheets will be analysed for omissions and missing data completed before being logged onto a central database and analysed by the research team at Imperial College, London, St. Mary's Campus.

The two groups will be compared using simple statistical methods. We intend to analyse and report on the following

* The number of patients who accepted inclusion into a pre-operative prehabilitation programme will be calculated.
* The change in physical fitness of patients (assessed by the physical function section of SF-36 and measured with peak flow/6-minute walk testing) during the pre-operative phase will be assessed pre and post-intervention groups.
* The effects on quality of life.
* The effect of a programme on anxiety and depression on each study participant will be assessed.
* The number of patients who are able to reduce or cease smoking will be reported.
* Compliance and acceptability of the prehabilitation programme.
* Morbidity and Mortality, HDU/ITU resource use as well as Length of hospital stay after aortic surgery.

ELIGIBILITY:
Inclusion Criteria:

- patients undergoing elective repair, willing/able to undertake a period of prehabilitation, and those able to comprehend and retain instructions regarding self-training.

Exclusion Criteria:

- Symptomatic patients or those undergoing urgent treatment (< 2 weeks)

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

IPD SHARING:
Plan to Share IPD: No
This trial did not complete as expected and therefore there are no meaningful participant data to share.

REFERENCES:
- [Background] Rooks DS, Huang J, Bierbaum BE, Bolus SA, Rubano J, Connolly CE, Alpert S, Iversen MD, Katz JN. Effect of preoperative exercise on measures of functional status in men and women undergoing total hip and knee arthroplasty. Arthritis Rheum. 2006 Oct 15;55(5):700-8. doi: 10.1002/art.22223. PMID 17013852
- [Background] Mayo NE, Feldman L, Scott S, Zavorsky G, Kim DJ, Charlebois P, Stein B, Carli F. Impact of preoperative change in physical function on postoperative recovery: argument supporting prehabilitation for colorectal surgery. Surgery. 2011 Sep;150(3):505-14. doi: 10.1016/j.surg.2011.07.045. PMID 21878237
- [Background] Kim DJ, Mayo NE, Carli F, Montgomery DL, Zavorsky GS. Responsive measures to prehabilitation in patients undergoing bowel resection surgery. Tohoku J Exp Med. 2009 Feb;217(2):109-15. doi: 10.1620/tjem.217.109. PMID 19212103
- [Background] Li C, Carli F, Lee L, Charlebois P, Stein B, Liberman AS, Kaneva P, Augustin B, Wongyingsinn M, Gamsa A, Kim DJ, Vassiliou MC, Feldman LS. Impact of a trimodal prehabilitation program on functional recovery after colorectal cancer surgery: a pilot study. Surg Endosc. 2013 Apr;27(4):1072-82. doi: 10.1007/s00464-012-2560-5. Epub 2012 Oct 9. PMID 23052535
- [Background] Carli F, Charlebois P, Stein B, Feldman L, Zavorsky G, Kim DJ, Scott S, Mayo NE. Randomized clinical trial of prehabilitation in colorectal surgery. Br J Surg. 2010 Aug;97(8):1187-97. doi: 10.1002/bjs.7102. PMID 20602503
- [Background] Dunckley M, Ellard D, Quinn T, Barlow J. Coronary artery bypass grafting: patients' and health professionals' views of recovery after hospital discharge. Eur J Cardiovasc Nurs. 2008 Mar;7(1):36-42. doi: 10.1016/j.ejcnurse.2007.06.001. Epub 2007 Jul 23. PMID 17644041
- [Background] Kiecolt-Glaser JK, Page GG, Marucha PT, MacCallum RC, Glaser R. Psychological influences on surgical recovery. Perspectives from psychoneuroimmunology. Am Psychol. 1998 Nov;53(11):1209-18. doi: 10.1037//0003-066x.53.11.1209. PMID 9830373
- [Background] Devine EC. Effects of psychoeducational care for adult surgical patients: a meta-analysis of 191 studies. Patient Educ Couns. 1992 Apr;19(2):129-42. doi: 10.1016/0738-3991(92)90193-m. PMID 1299818
- [Background] Mumford E, Schlesinger HJ, Glass GV. The effect of psychological intervention on recovery from surgery and heart attacks: an analysis of the literature. Am J Public Health. 1982 Feb;72(2):141-51. doi: 10.2105/ajph.72.2.141. PMID 7055315
- [Background] Furze G, Dumville JC, Miles JN, Irvine K, Thompson DR, Lewin RJ. "Prehabilitation" prior to CABG surgery improves physical functioning and depression. Int J Cardiol. 2009 Feb 6;132(1):51-8. doi: 10.1016/j.ijcard.2008.06.001. Epub 2008 Aug 15. PMID 18703241
- [Background] Owen D, Bicknell C, Hilton C, Lind J, Jalloh I, Owen M, Harrison R. Preoperative smoking cessation: a questionnaire study. Int J Clin Pract. 2007 Dec;61(12):2002-4. doi: 10.1111/j.1742-1241.2007.01565..x. Epub 2007 Sep 10. PMID 17850308
- [Background] Arthur HM, Daniels C, McKelvie R, Hirsh J, Rush B. Effect of a preoperative intervention on preoperative and postoperative outcomes in low-risk patients awaiting elective coronary artery bypass graft surgery. A randomized, controlled trial. Ann Intern Med. 2000 Aug 15;133(4):253-62. doi: 10.7326/0003-4819-133-4-200008150-00007. PMID 10929164
- [Background] Cunningham MA, Swanson V, O'Carroll RE, Holdsworth RJ. Randomized clinical trial of a brief psychological intervention to increase walking in patients with intermittent claudication. Br J Surg. 2012 Jan;99(1):49-56. doi: 10.1002/bjs.7714. Epub 2011 Oct 28. PMID 22038532
- [Background] Hlatky MA, Boineau RE, Higginbotham MB, Lee KL, Mark DB, Califf RM, Cobb FR, Pryor DB. A brief self-administered questionnaire to determine functional capacity (the Duke Activity Status Index). Am J Cardiol. 1989 Sep 15;64(10):651-4. doi: 10.1016/0002-9149(89)90496-7. PMID 2782256

RESULTS

PARTICIPANT FLOW:
Groups:
- Post-intervention: Patients after the institution of a physical, psychological and social training programme
  Prehabilitation: Introduction of a physical exercise training programme, psychological counselling and smoking cessation advice
Period: Overall Study
Arm/Group | Pre-intervention | Post-intervention
Started | 13 | 12
Completed | 0 | 5
Not Completed | 13 | 7
Not completed — Protocol Violation | 13 | 7

BASELINE CHARACTERISTICS:
Groups:
- Baseline Pre: Baseline Characteristics of the Pre-intervention Standard of Care
- Baseline Post: Baseline Characteristics of the Post-intervention Prehabilitation
- Total: Total of all reporting groups
Arm/Group | Baseline Pre | Baseline Post | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 11 | 9 | 20
Age, Continuous [Mean (Full Range); unit: years] | 74.3 [60 to 87] | 70.8 [49 to 83] | 72.64 [49 to 87]
Sex/Gender, Customized [Number; unit: participants]
  Female | 2 | 3 | 5
  Male | 11 | 9 | 20
Region of Enrollment [Number; unit: participants] — Imperial Vascular Unit
  participants
    United Kingdom | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients Who Accepted Inclusion Into a Pre-operative Prehabilitation Programme
Description: This describes the number of people within the study who were in the pre-habilitation study arm that accepted and completed the pre-habilitation training
Time Frame: Collected at screening
Measure: Number; unit: participants
Arm/Group | Post-intervention
Number analyzed (Participants) | 12
participants | 11

2. Primary Outcome: Change From Baseline in Metabolic Equivalents (METS) at Six Weeks
Description: • Metabolic equivalent level is a measure of physical fitness. One MET is defined as 3.5 mL 02 uptake/kg per minute which is the resting oxygen uptake in a sitting position. The achieved exercise capacity in METs has been shown to be predictive in older adult population of survival with higher MET levels associated with improved survival," or similar definition that is accurate and appropriate.
Time Frame: Collected at baseline and (expected) 6 weeks
Population: There were no patients in the pre-intervention group who underwent pre-operative METS testing
Measure: Mean (Full Range); unit: METS
Groups:
- Pre-intervention: Before the introduction of a rehabilitation programme
Arm/Group | Post-intervention | Pre-intervention
Number analyzed (Participants) | 5 | 0
METS | 0.06 [0 to 0.1] |

3. Primary Outcome: Decrease in Anxiety and Depression Scores (Hospital Anxiety and Depression Scale)
Description: HADS is a validated questionnaire consisting of 7 statements relating to anxiety and 7 statements relating to depression. Each statement is scored between 0 and 3 giving a total score of up to 21 for each section. A score of 0-7 is assumed to be normal and score greater than this suggestive of a mood disorder
Time Frame: Collected at baseline and (expected) 6 weeks
Population: There were no patients in the pre-intervention group who underwent pre-operative HADS testing
Measure: Mean (Full Range); unit: HADS scores
Groups:
- Pre-intervention: Before the institution of a rehabilitation programme
Arm/Group | Post-intervention | Pre-intervention
Number analyzed (Participants) | 5 | 0
HADS scores
  HADS - D | 1.2 [-3 to 4] |
  HADS - A | 5 [-2 to 9] |

4. Primary Outcome: Number of Participants With Attendance at the Physical and Psychological and Social Training Appointments of the Rehabilitation Programme (Assessed by Bespoke Questionnaire)
Time Frame: Collected at baseline and during the study
Measure: Count of Participants; unit: Participants
Arm/Group | Post-intervention
Number analyzed (Participants) | 12
Participants | 11

5. Secondary Outcome: HDU/ITU Resource Use (Number of Days Stay)
Description: Observation to power a larger intervention study
Time Frame: Collected at (expected) 6 weeks +hospital stay
Population: The number of participants where post operative HDU/ITU stay information was available was significantly reduced as this information was not collected by the study reporting team.
Measure: Mean (Full Range); unit: Days
Groups:
- Post-intervention: Patients after the institution of a physical, psychological and social training programme
  Prehabilitation: Introduction of a physical exercise training programme, psychological counselling and smoking cessation advice = 13
Arm/Group | Pre-intervention | Post-intervention
Number analyzed (Participants) | 4 | 7
Days | 1.75 [1 to 3] | 2.42 [1 to 5]

6. Secondary Outcome: LOS
Description: Length of hospital stay after aortic surgery (number of days) - Observation to power a larger intervention study
Time Frame: Collected at (expected) 6 weeks +hospital stay
Population: The number of participants where length of hospital stay information was available was significantly reduced as this information was not collected by the study reporting team.
Measure: Mean (Full Range); unit: days
Arm/Group | Pre-intervention | Post-intervention
Number analyzed (Participants) | 7 | 4
days | 5.5 [4 to 8] | 5.14 [2 to 7]

ADVERSE EVENTS:
Groups:
- Pre-intervention: Before the institution of a physical, psychological and social training programme
Arm/Group | Post-intervention | Pre-intervention
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13

LIMITATIONS AND CAVEATS:
There was a significant failure in patients undergoing METS and HADS assessment prior to surgery and therefore the results of this pilot study are limited to a lot study of whether patients accepted this intensive rehabilitation study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes